CLINICAL TRIAL: NCT02251223
Title: An Open Label Multinational Study of the Effects of Three Dose Pairs of Tipranavir/Ritonavir (b.i.d.) on the Pharmacokinetic Characteristics of Protocol -Defined, Baseline, Triple Drug Nucleoside and Non-nucleoside Reverse Transcriptase Inhibitor Therapy in HIV-1-infected Subjects.
Brief Title: Effects of Tipranavir/Ritonavir on the Pharmacokinetic Characteristics of Triple Drug Nucleoside and Non-nucleoside Reverse Transcriptase Inhibitor Therapy in HIV-1-infected Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 1182.6
Record Dates: First submitted 2014-09-25; First posted 2014-09-29 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-09

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — tipranavir; Ritonavir

ARMS (3):
- TPV/r low dose (Experimental)
  Interventions: Drug: Tipranavir low dose; Drug: Ritonavir high dose
- TPV/r medium dose (Experimental)
  Interventions: Drug: Tipranavir medium dose; Drug: Ritonavir low dose
- TPV/r high dose (Experimental)
  Interventions: Drug: Tipranavir high dose; Drug: Ritonavir low dose

INTERVENTIONS:
Drug: Tipranavir low dose
  Arms: TPV/r low dose
Drug: Tipranavir medium dose
  Arms: TPV/r medium dose
Drug: Tipranavir high dose
  Arms: TPV/r high dose
Drug: Ritonavir low dose
  Arms: TPV/r high dose; TPV/r medium dose
Drug: Ritonavir high dose
  Arms: TPV/r low dose

SUMMARY:
Primary: Sequentially determine the effects of three dose combinations of tipranavir (TPV) / ritonavir (RTV) (administered b.i.d.), TPV 1250 mg/RTV 100 mg vs. TPV 750 mg/RTV 100 mg vs. TPV 250 mg/RTV 200 mg on the steady-state pharmacokinetics of zidovudine, lamivudine, stavudine, didanosine, abacavir, nevirapine and efavirenz at approved doses. The three treatment groups will be enrolled sequentially starting with the highest tipranavir dosage group first and ending with the lowest tipranavir dosage group.

Secondary: A) To assess the effects of zidovudine, lamivudine, stavudine, didanosine, abacavir, nevirapine, and efavirenz on the pharmacokinetics of tipranavir/ritonavir compared to historical controls.

B) To assess the safety of three tipranavir/ritonavir combinations when used in combination with protocol defined antiretrovirals.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent prior to trial participation
2. Between 18 and 75 years of age inclusive
3. Female subjects of child bearing potential are required to use a barrier contraceptive method for at least 12 weeks prior to administration of study medication, during study medication administration, and for 28 days after the end of the study
4. Ability to swallow capsules without difficulty
5. A Body Mass Index (BMI) between 11 and 50 kg/m2
6. Reasonable probability for completion of the study
7. Acceptable screening laboratory values. All laboratory values ≤ Grade I (e.g., creatine phosphokinase (CPK), amylase, triglycerides) are permissible if documentation of stability for 2 months or more is available. Abnormalities > Grade I are subject to approval by BI clinical monitor or designee
8. Acceptable medical history, physical examination, ECG, and chest X-ray prior to entering the treatment phase of the study
9. Willingness to abstain from alcohol from Day -2 to Day 23
10. Willingness to abstain from ingesting grapefruit, grapefruit juice, Seville oranges or orange marmalade from Day -2 to Day 23
11. Negative urine drug screen for drugs of abuse. Subjects on methadone or equivalent narcotic maintenance programs will be permitted to enter the study
12. Documented HIV-1 RNA load (by PCR) at screening of ≤20,000 copies/mL for at least twelve weeks. Acceptable documentation would include laboratory data, a letter or a verbal report from another provider noted in the subject records.
13. Stable doses of approved NRTIs and NNRTIs 2 for a minimum of twelve weeks prior to study Day 0. Subjects on efavirenz must be able to tolerate daily morning (8:00 a.m.) dosing starting at screening period and for 22 days of the study. Subjects receiving bid ddI must be willing to accept a change to the once a day delayed release (EC) formulation

Exclusion Criteria:

1. Female subjects who:

   * have a positive serum pregnancy test at Screening Period Day -14 to -7
   * are breast feeding
2. Receipt of any other investigational medicine for 30 days prior to Day 0
3. Receipt of any known cytochrome P450 3A4 (CYP3A4) altering drug i.e. phenothiazines, cimetidine, barbiturates, ketoconazole, fluconazole, rifampin, steroids and herbal medications for 30 days prior to Day 0. No antibiotics permitted within 10 days prior to Day 0
4. Ingestion of grapefruit, grapefruit juice, Seville oranges or orange marmalade within 2 days of study entry (Day 0)
5. Blood or plasma donations (>100 ml total) for research or altruistic reasons within 30 days prior to Day 0
6. Seated systolic blood pressure either <100 mm Hg or >150 mm Hg; resting heart rate either <50 beats/minute or >90 beats/minute
7. History of any illness, including malabsorption, irregular food intake or gastrointestinal intolerance, or allergy that, in the opinion of the investigator, might confound the results of the study or pose additional risk in administering TPV/RTV
8. Any acute illness within 2 weeks prior to Day 0
9. Subjects who are currently taking any over-the-counter drug within 7 days prior to Day 0, or who are currently taking any prescription drug that, in the opinion of the investigator (in consultation with the BI medical monitor and/or pharmacokineticist), might interfere with either the absorption, distribution or metabolism of the TPV/RTV
10. Hypersensitivity to TPV, RTV or sulfonamide containing drugs
11. Using the adherence diary, subject has less than 100% documented adherence for the last 14 doses (7 days) of baseline antiretroviral medications prior to Day 0. Subjects has less than 100% adherence for the last 7 doses (7 days) of efavirenz and ddI (delayed release) prior to Day 0

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2001-02; Primary Completion 2002-02 (Actual)

PRIMARY OUTCOMES:
Change in trough plasma concentration (Cmin,ss) for non-nucleoside reverse transcriptase inhibitor (NNRTI) | baseline, up to day 23
  stratified by substance
Change in area under plasma concentration-time curve over dosing interval (AUC0-τ) for nucleoside reverse transcriptase inhibitor (NRTI) | baseline, up to day 22
  stratified by substance
Change in area under plasma concentration-time curve from 0 to 12 hours for didanosine (ddI) | baseline, up to day 22

SECONDARY OUTCOMES:
Cmin,ss | up to day 23
  stratified by substance
AUC0-τ | up to day 23
  stratified by substance
Maximum plasma concentration (Cmax) | up to day 23
  stratified by substance
Time of maximum plasma concentration (Tmax) | up to day 23
  stratified by substance
Oral clearance (Cl/F) | up to day 23
  stratified by substance
Apparent terminal half life (t1/2) | up to day 23
  stratified by substance
Change in CD4 cell count | up to day 23
Change in HIV-1 RNA levels | up to day 23
Number of patients with clinically significant findings in laboratory tests | up to 25 weeks
Number of patients with adverse events | up to 25 weeks